CLINICAL TRIAL: NCT00197262
Title: A Randomized, Single-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy of Once-Daily, Intranasal Administration of GW685698X Aqueous Nasal Spray 100 mcg for 2 Weeks in Adult and Adolescent Subjects With Seasonal Allergic Rhinitis
Brief Title: Once-Daily Investigational Nasal Spray In Adults And Adolescents With Seasonal Allergic Rhinitis (SAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR104861
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Seasonal Allergic Rhinitis; GW685698X; allergic rhinitis; Hayfever
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW685698X Aqueous Nasal Spray

SUMMARY:
Allergic rhinitis is an inflammatory disorder of the upper airway that occurs following allergen exposure. The focus of this study, seasonal allergic rhinitis (SAR), is one type of allergic rhinitis that is triggered by the pollen from trees, grasses, and weeds. Commonly referred to as (hay fever), it is characterized by sneezing, nasal congestion and pruritus, rhinorrhea, and pruritic, watery, red eyes. The primary objective of this study is to compare the efficacy and safety of GW685698X 100mcg once daily (QD) aqueous nasal spray with vehicle placebo nasal spray in adult and adolescent subjects (12 years of age and older) with seasonal allergic rhinitis (SAR) caused by ragweed pollen.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Once-Daily, Intranasal Administration of GW685698X Aqueous Nasal Spray 100mcg for 2 Weeks in Adult and Adolescent Subjects (12 years of age and older) with Seasonal Allergic Rhinitis (SAR)

ELIGIBILITY:
Inclusion criteria:

* Must be outpatients.
* Diagnosis of SAR.
* Literate in English or native language.

Exclusion criteria:

* Have a significant concomitant medical condition.
* Use corticosteroids or other allergy medications during the study.
* Use tobacco products.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288
Dates: Start 2005-08; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline over the entire treatment period in daily, reflective total nasal symptom scores.

SECONDARY OUTCOMES:
1) Mean change from baseline over the entire treatment period in AM, pre-dose, instantaneous total nasal symptom scores. 2) Mean change from baseline in daily reflective total ocular symptom scores. 3) overall evaluation of response to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- United States (17):
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Novi, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Greenfield, Wisconsin
  - GSK Investigational Site, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: FFR104861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR104861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR104861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR104861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR104861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR104861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR104861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register